CLINICAL TRIAL: NCT01397799
Title: A Phase 1b Rising Multiple-Dose Study to Evaluate Safety, Tolerability and Activity of KX2-391 in Elderly Subjects With Acute Myeloid Leukemia Who Are Refractory to or Have Declined Standard Induction Therapy
Brief Title: Evaluation of KX2-391 in Elderly Subjects With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kinex Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Organization: Athenex, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX01-03-11
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Acute Myelogenous Leukemia; AML; Refractory; Elderly
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tirbanibulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Subjects will be enrolled into a 28-day dose-escalation study. If no DLT's are observed during the first 28 days, subjects are eligible to continue treatment in the Extension Phase and can remain on treatment until toxicity occurs or until disease progression.
  Interventions: Drug: KX2-391

INTERVENTIONS:
Drug: KX2-391 — Oral dose solution, once-daily dosing for 28-days. Subjects may continue beyond the first 28-days until disease progression or unacceptable toxicity develops.
  Other Names: KX01

SUMMARY:
This Phase 1b study will determine the maximum tolerated dose of KX2-391 given as a once-daily dose, in elderly patients with acute myelogenous leukemia.

DETAILED DESCRIPTION:
KX2-391 has been evaluated in a Phase 1 dose escalation study in patients with solid tumors using twice-daily dosing. This study will employ the Storer's two-stage design to determine the maximum tolerated dose of KX2-391 mono-therapy,given as a once-daily oral dose,in elderly patients with acute myelogenous leukemia (AML) who are refractory to or have declined standard induction therapy. The safety, tolerability, pharmacokinetics and activity of KX2-391 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Either de novo or secondary AML by 2008 World Health Organization (WHO) classification.
* A bone marrow biopsy and aspirate sample must be obtained between Day -14 to Day -1, and this sample must be confirmed to be adequate for morphologic analysis of marrow cellularity and blast percentage before the first dose of KX2-391 is administered.
* A bone aspirate sample (with or without biopsy) must be obtained after the patient signs the informed consent document and be submitted for baseline pharmacodynamic assessment. Although this will usually be obtained as part of the baseline assessment marrow biopsy and aspirate procedure described above, if a complete marrow evaluation was performed prior to the patient signing informed consent, a dedicated bone marrow aspiration for this sample can be performed after the patient signs informed consent, so long as the pre-consent biopsy and aspirate procedure were done within 14 days of the first dose of KX2-391.
* Adults age ≥ 60 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Life expectancy of at least 6 weeks from first day of study drug administration
* Adequate liver function (AST/ALT < 3 x upper limit of normal (ULN), Alk Phos < 2.5 x ULN, and Direct Bilirubin < 1.5 x ULN)
* Adequate renal function (serum creatinine < 1.5 x ULN)
* Documented QTc ≤ 0.48 seconds within 14 days of first dose of KX2-391

Exclusion Criteria:

* Subjects with acute promyelocytic leukemia (APL, AML FAB type M3), or chronic myelogenous leukemia (CML).
* Have not resolved toxicity from previous anticancer treatments or investigational agents, other than hematologic toxicities or alopecia, to ≤ Grade 1 according to the most recent CTCAE guidelines.
* Subjects with rapidly proliferative AML that is likely to require treatment within the next 30 days (e.g. hydroxyurea).
* Received an investigational agent within 5 half-lives of that agent from the anticipated Cycle 1 Day 1 of treatment with KX2-391.
* Have clinical evidence of central nervous system involvement by AML or other malignancy.
* History of major surgery to the upper gastrointestinal tract, or have a history of inflammatory bowel disease, malabsorption syndrome, or other medical condition that may interfere with oral drug absorption.
* Uncontrolled hypertension (at time of dosing).
* Other medical conditions which, in the opinion of the investigator, make it undesirable for the subject to participate in the study.
* Known history of hepatitis B, C, or human immunodeficiency (HIV) infection.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection. Patients receiving intravenous antibiotics for infections that are under control may be included in this study.
* Subjects who are unwilling or unable to comply with the protocol.
* Subjects who are taking moderate or strong CYP450 3A4 modulators, with the exception of fluconazole (see Appendix 2 for list of medications currently known to be moderate or strong CYP450 3A4 modulators). Subjects who can safely discontinue these medications can become eligible for this trial.
* Subjects receiving azole-based antifungal prophylaxis other than fluconazole (see Appendix 2) who are unable to switch their prophylaxis to fluconazole, or discontinue antifungal prophylaxis, for 7 days prior to first day of study drug administration.
* Active cancer, other than AML, requiring systemic chemotherapy or biological therapy within 6 months of study entry. Patients who have received only hormonal therapy in the neoadjuvant or adjuvant setting in the past 6 months may participate in this study.
* Symptomatic congestive heart failure, unstable angina, or cardiac arrhythmia.
* Other conditions that could jeopardize the subject's ability to comply with the protocol, including, but not limited to, dementia, psychosis, or other major psychiatric disorder
* Pregnant or breast feeding

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of KX2-391 when given once-daily to AML patients. | 28 days
  The MTD will be used to determine the recommended Phase 2 dose that is associated with an approximately 33% DLT rate during the first 28 days of treatment in elderly patients with AML

SECONDARY OUTCOMES:
Evaluate pharmacokinetics, pharmacodynamics and activity of KX2-391. | 28 days
  The pharmacokinetics and pharmacodynamics of KX2-391 will be evaluated in AML patients by measuring serum and bone marrow levels of drug and evaluating the disruption of microtubule networks in these samples to determine whether target inhibition has occurred at the doses tested. Hematological and bone marrow response will be assessed according to International Working Group (IWG)-AML criteria.

CONTACTS AND LOCATIONS:
Overall Officials: James Thompson, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (3):
- United States (3):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Kasner MT, Halloran MB, Pan J, Ritchie EK, Fetterly GJ, Kramer D, Hangauer DG, Thompson JE. A phase Ib dose escalation study of oral monotherapy with KX2-391 in elderly patients with acute myeloid leukemia. Invest New Drugs. 2022 Aug;40(4):773-781. doi: 10.1007/s10637-022-01255-1. Epub 2022 May 17. PMID 35579731